CLINICAL TRIAL: NCT00707369
Title: Adjunctive Antimicrobial Therapy of Periodontitis: Long-Term Effects on Disease Progression and Oral Microbiological Colonization
Acronym: ABPARO-Studie
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Benjamin Ehmke, Prof. Dr. med. dent., University Hospital Muenster
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EH 365/1-1; DFG grant: EH 365/1-1; ISRCTN : 64254080
Record Dates: First submitted 2008-06-24; First posted 2008-06-30 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Periodontitis
Keywords: Periodontitis; Mechanical Debridement; Antibiotics; Attachment loss; Randomized controlled trial
MeSH Terms: conditions — Periodontitis | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- test (Experimental): Mechanical debridement plus 500 mg amoxicillin and 400 mg metronidazole three times daily for 7 days. Supportive periodontal therapy in 3-month intervals.
  Interventions: Drug: Amoxicillin and Metronidazole
- control (Placebo Comparator): Mechanical debridement plus two placebo tablets three times daily for 7 days. Supportive periodontal therapy in 3-month intervals.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amoxicillin and Metronidazole — tablets: Amoxicillin 3H2O 574 mg and 400 mg metronidazole three times daily for 7 days
  Other Names: Flagyl® 400 Filmtablette; Amoxicillin-ratiopharm® 500
  Arms: test
Drug: Placebo — Placebo tablets (cellulose powder, lactose monohydrate, magnesium stearate, microcrystalline cellulose): three times daily for 7 days
  Arms: control

SUMMARY:
The purpose of this study is to determine the size of the benefit of an adjunctive empiric antibiotic therapy compared to standard mechanical debridement and oral hygiene instructions in a representative sample of German periodontitis patients.

DETAILED DESCRIPTION:
Periodontitis is an endemic inflammatory disease caused by a mixed bacterial biofilm infection that is followed by destruction of tooth supporting tissues. Standard of care consists of lifelong mechanical removal of the biofilm. However, outcome is variable. According to recent EFP and AAP reviews, adjunctive antimicrobial therapy may be beneficial. We plan to conduct a double-blind, parallel group, randomized, placebo-controlled multi-center efficacy study that addresses the following objectives:

1. What is the size of the benefit of an adjunctive empiric antibiotic therapy compared to standard mechanical debridement and oral hygiene instructions in a representative sample of German periodontitis patients?
2. Does the administration of the antibiotic therapy delay recurrence of periodontitis in the general population and in specific high risk groups (e.g. smokers) under standard supportive therapy?
3. Is the presence of specific microbial complexes a useful predictor of outcome and recurrence of periodontitis?
4. Does the administration of the antibiotic therapy affect the "oral health related quality of life"?

The primary hypothesis tested is: the administered empiric adjunctive antibiotic therapy reduces about one half of the proportion of sites with attachment loss compared to subgingival debridement alone over a 27.5-month period in a statistical and clinical significant manner.

To test this hypothesis about 500 patients will be enrolled in the clinical trial. According to the intention-to-treat principle, the primary efficacy analysis will include all randomized subjects. In addition, a per-protocol analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* periodontal screening index (PSI) of IV in at least one sextant;
* range from 18 to 75 years of age;
* clinical and radiographic signs of moderate (clinical attachment loss [CAL] of 3 to 4 mm) to severe (CAL 5 mm or more) chronic or aggressive periodontitis;
* at least 10 natural teeth in situ;
* pocket probing depths (PPDs) of ≥ 6 mm at a minimum of four teeth;
* willingness to participate and to be available at all times required for participation;
* willingness to abstain from using antimicrobial mouth-rinses during the study except for those explicitly prescribed;
* informed consent signed by the patient;
* sufficient knowledge of German language.

Exclusion Criteria:

* if they (or parents or siblings) show confirmed or assumed allergies or hyper-sensitive skin reactions against amoxicillin (or other penicillins or other ingredients of Amoxicillin-ratiopharm® 500mg as listed in the "summary of product characteristics, Version Juli 2005"), metronidazole (or other 5-nitroimidazoles and ingredients of Flagyl® 400mg as listed in the "summary of product characteristics, Version Juli 2007"), systemic diseases or conditions as listed in the above mentioned "summary of product characteristics", or show confirmed lactose intolerance;
* have Down's syndrome;
* known AIDS/HIV;
* regularly take systemic medication affecting the periodontal conditions, e.g. phenytoin, nifedipine, and/or steroid drugs;
* professional periodontal therapy during 6 months prior to baseline;
* require antibiotic treatment for dental appointments;
* are undergoing or require extensive dental or orthodontic treatment;
* are pregnant or breastfeeding;
* have rampant caries;
* any oral or extraoral piercing in or around the oral cavity with ornaments or accessory jewelry;
* are dental students or dental professionals;
* have participated in a clinical dental trial in the six months preceding the study;
* cognitive deficits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Percentage of sites showing attachment loss ≥ 1.3 mm over a 27.5-months period | 27.5-months period (six measurements)

SECONDARY OUTCOMES:
Subjective perception of treatment outcome, attachment gain, pocket probing depths, bleeding on probing, and full mouth plaque score. Microbial colonization dynamic. | over a 27.5-months period

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin - Ehmke, PhD, Principal Investigator — University Hospital Muenster, Dept. of Periodontology
Locations (8):
- Germany (8):
  - Medizinische Fakultät der Humboldt Universität Berlin (Charité), Berlin
  - Universitätsklinikum Carl Gustav Carus, Zentrum für Zahn-, Mund- und Kieferheilkunde, Dresden
  - Zentrum der Zahn-, Mund- und Kieferheilkunde (Carolinum), Poliklinik für Parodontologie, Frankfurt
  - Justus-Liebig-Universität Gießen, Poliklinik für Parodontologie, Giessen
  - Universitätsklinikum Greifswald, Poliklinik für Zahnerhaltung, Parodontologie und Kinderzahnheilkunde, Greifswald
  - Universitätsklinikum Heidelberg, Poliklinik für Zahnerhaltungskunde, Sektion Parodontologie, Heidelberg
  - University Hospital Muenster, Dept. of Periodontology, Münster
  - Universität Würzburg, Poliklinik für Parodontologie, Würzburg

REFERENCES:
- [Derived] Walther KA, Gonzales JR, Groger S, Ehmke B, Kaner D, Lorenz K, Eickholz P, Kocher T, Kim TS, Schlagenhauf U, Koch R, Meyle J. The Role of Polymorphisms at the Interleukin-1, Interleukin-4, GATA-3 and Cyclooxygenase-2 Genes in Non-Surgical Periodontal Therapy. Int J Mol Sci. 2022 Jun 30;23(13):7266. doi: 10.3390/ijms23137266. PMID 35806269
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289
- [Derived] Matern J, Koch R, Petersmann A, Kocher T, Eickholz P, Lorenz K, Kim TS, Meyle J, Kaner D, Schlagenhauf U, Gravemeier M, Harks I, Ehmke B. Effect of periodontal therapy on adipokine biomarkers in overweight. J Clin Periodontol. 2020 Jul;47(7):842-850. doi: 10.1111/jcpe.13288. Epub 2020 May 11. PMID 32248552
- [Derived] Eickholz P, Koch R, Kocher T, Hoffmann T, Kim TS, Meyle J, Kaner D, Schlagenhauf U, Harmsen D, Harks I, Ehmke B. Clinical benefits of systemic amoxicillin/metronidazole may depend on periodontitis severity and patients' age: An exploratory sub-analysis of the ABPARO trial. J Clin Periodontol. 2019 Apr;46(4):491-501. doi: 10.1111/jcpe.13096. Epub 2019 Apr 12. PMID 30825384
- [Derived] Kocher T, Holtfreter B, Petersmann A, Eickholz P, Hoffmann T, Kaner D, Kim TS, Meyle J, Schlagenhauf U, Doering S, Gravemeier M, Prior K, Rathmann W, Harks I, Ehmke B, Koch R. Effect of Periodontal Treatment on HbA1c among Patients with Prediabetes. J Dent Res. 2019 Feb;98(2):171-179. doi: 10.1177/0022034518804185. Epub 2018 Oct 16. PMID 30326764
- [Derived] Eickholz P, Nickles K, Koch R, Harks I, Hoffmann T, Kim TS, Kocher T, Meyle J, Kaner D, Schlagenhauf U, Doering S, Gravemeier M, Ehmke B. Is furcation involvement affected by adjunctive systemic amoxicillin plus metronidazole? A clinical trials exploratory subanalysis. J Clin Periodontol. 2016 Oct;43(10):839-48. doi: 10.1111/jcpe.12594. Epub 2016 Aug 10. PMID 27393928
- [Derived] Harks I, Koch R, Eickholz P, Hoffmann T, Kim TS, Kocher T, Meyle J, Kaner D, Schlagenhauf U, Doering S, Holtfreter B, Gravemeier M, Harmsen D, Ehmke B. Is progression of periodontitis relevantly influenced by systemic antibiotics? A clinical randomized trial. J Clin Periodontol. 2015 Sep;42(9):832-842. doi: 10.1111/jcpe.12441. Epub 2015 Sep 22. PMID 26250060